CLINICAL TRIAL: NCT05162807
Title: Improving Caregiver Palliative Care Knowledge and Attitudes: Evaluating the Impact of a Psychoeducational Intervention
Brief Title: Intervention to Improve Caregiver Palliative Care Knowledge and Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Brenna K Mossman, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1041
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cancer
Keywords: Palliative care; Caregiver
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Between groups, randomized design. Participants are randomized to either intervention or control conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Education (Experimental): The intervention arm will view a psychoeducational video on palliative care.
  Interventions: Behavioral: Psychoeducational Video on Palliative Care
- Attention Control (Placebo Comparator): The control arm will view an educational video on nutrition as an attention control.
  Interventions: Behavioral: Educational Video on Nutrition

INTERVENTIONS:
Behavioral: Psychoeducational Video on Palliative Care — The intervention is a psychoeducational video introducing palliative care and discussing its purpose, structure, benefits, and efficacy.
  Arms: Palliative Care Education
Behavioral: Educational Video on Nutrition — The attention control is a video on nutrition and healthy eating during cancer survivorship.
  Arms: Attention Control

SUMMARY:
This randomized clinical trial will assess whether a psychoeducational intervention will improve palliative care knowledge and attitudes among close friends and family members of individuals with cancer. The psychoeducational intervention entails viewing a video introducing palliative care and its purpose, structure, benefits, and efficacy.

DETAILED DESCRIPTION:
The primary aims of this randomized clinical trial are to examine the impact of a psychoeducational intervention on (1) palliative care knowledge, and (2) palliative care attitudes among close friends and family members of individuals with cancer. Participants will complete a baseline survey including measures of palliative care knowledge and experience. Participants will be randomized to then view either a psychoeducational video introducing palliative care (intervention) or an educational video on nutrition throughout cancer survivorship (attention control). All participants will then complete outcome measures, including primary outcomes of palliative care knowledge and attitudes.

ELIGIBILITY:
Inclusion criteria:

* Provide informed consent
* 18 years of age or older
* Have ever had a close friend or family member diagnosed with cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Palliative Care Knowledge Scale (PaCKS) | Immediately post-intervention
  Participants in both groups will complete the 13-item Palliative Care Knowledge Scale (PaCKS). The scale presents a series of items about palliative care, and response options reflect whether participants believe the items are true or false, or whether the participant does not know the answer. Each correct answer will be scored as 1, each incorrect or unsure answer will be scored as 0, and correct responses will be summed to create a total score. The total score will range from 0-13, with higher scores indicating greater palliative care knowledge.
Palliative Care Attitudes Scale - Caregiver (PCAS-9C) | Immediately post-intervention
  Participants in both groups will report attitudes toward palliative care by completing the 9-item Palliative Care Attitudes Scale for Caregivers (PCAS-9C). The PCAS-9C consists of three subscales with three items each: emotional (reverse-coded), cognitive, and behavioral. Participants rate each item from 1 to 5. Total scores will range from 9 to 45, with higher scores indicating more favorable attitudes towards palliative care.

CONTACTS AND LOCATIONS:
Overall Officials: Brenna K Mossman, MA, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States